CLINICAL TRIAL: NCT06090422
Title: Ketamine for Combined Depression and Alcohol Use Disorder: A Blinded Randomized Active Placebo-controlled Trial (the KeDA Trial)
Brief Title: Ketamine for Combined Depression and Alcohol Use Disorder
Acronym: KeDA
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Principal Investigator, Andreas Wahl Blomkvist, Principal Investigator, University Hospital of North Norway
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022/484848(REK); 2023-506052-24 (EudraCT Number); U1111-1293-2654 (Other: WHO UTN)
Record Dates: First submitted 2023-07-01; First posted 2023-10-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Depression; Alcohol Use Disorder
Keywords: Depression; Alcohol use disorder; Ketamine; Addiction
MeSH Terms: conditions — Depression; Alcoholism; Behavior, Addictive | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Ketamine, 0,8 mg/kg body weight, given as four single doses (biweekly for two weeks)
  Interventions: Drug: Ketamine Hydrochloride
- Control group (Active Comparator): Midazolam, 0,8 mg/kg body weight, given as four single doses (biweekly for two weeks)
  Interventions: Drug: Midazolam Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Four single-doses, given two times per week for two weeks Dose: 0,8 mg/kg body weight Route of administration: intravenous infusions over 40 minutes
  Arms: Intervention group
Drug: Midazolam Hydrochloride — Four single-doses, given two times per week for two weeks Dose: 0,02 mg/kg body weight Route of administration: intravenous infusions over 40 minutes
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to investigate the effects of ketamine, in combination with standard inpatient addiction therapy, for adults with depression and alcohol use disorder. After screening and enrollment, participants will undergo baseline assessments of depression, measures of alcohol use and craving, as well as neurocognitive function. Participants will then be randomized to either ketamine (intervention) or midazolam (control). All participants will be admitted for standard inpatient addiction therapy while receiving ketamine or midazolam. Measures on safety, depression and alcohol use disorder will be repeatedly assessed during and after treatment. Final follow-up assessment is scheduled 6 months after baseline assessment.

DETAILED DESCRIPTION:
Depression and alcohol use disorder (AUD) often coexist and can create significant challenges for individuals seeking effective treatment. Traditional treatment approaches have shown limited success in addressing both conditions simultaneously. Ketamine has shown to have promising rapid antidepressant effects and a possible role in the treatment of substance use disorders. By targeting both depression and AUD simultaneously, ketamine has the potential to offer dual benefits, improving depressive symptoms while addressing alcohol cravings or consumption. Furthermore, rapid relief from depressive symptoms may enhance motivation for recovery, reduce the risk of relapse, and improve overall treatment engagement and outcomes. Although ketamine is generally considered safe when administered under medical supervision, the safety profile in individuals with comorbid depression and AUD needs further investigation. The overall objective of this study is to examine the safety and efficacy of ketamine on adults with depression and AUD that are admitted for standard inpatient addiction therapy.

The study will only include adults with at least moderate depression and alcohol use disorder as their primary substance use disorder that are admitted for inpatient addiction therapy. Participants that are unable to give informed consent or have contraindication(s) for ketamine will be excluded.

After screening and enrollment, participants will undergo baseline assessments with measures on depression (using Montgomery-Åsberg Depression Rating Scale (MADRS) and Beck Depression Inventory-II (BDI-II)), alcohol use (using Timeline Follow-Back method (TLFB)), alcohol craving (using Short version of Alcohol Craving Questionnaire (ACQ-Short) and Penn Alcohol Craving Scale (PACS)) and neurocognitive function (using Cambridge Neuropsychological Test Automated Battery (CANTAB)). Participants will then be randomized to intervention group or control group. The intervention group will receive ketamine as four single doses, given biweekly for two weeks. The control group will receive midazolam as active placebo. Participants will undergo several follow-up assessments after treatment (1-2 day(s), 1 week, 2 weeks and 4 weeks after treatment). Final follow-up assessment will be 6 months after baseline.

By using open questions and specific instruments for assessing adverse effects associated with ketamine (using modified version of Ketamine Side Effect Tool (mKSET)), the trial will assess the frequency, severity and duration of any adverse events and severe adverse events. All adverse events will be evaluated with regards to its causal relationship to ketamine. In addition, physician-assessed and patient-assessed tolerability will be registered. Changes in neurocognitive function from baseline will be assessed after treatment.

Changes in depression will be measured several times using rater-blinded MADRS-assessment and self-report instrument (BDI-II). Measures of alcohol use (TLFB), alcohol craving (ACQ-short and PACS), relapse risk and time until relapse will used as measures on alcohol use disorder following treatment. Several exploratory objectives will be examined, including changes in alcohol dependence severity (using Severity of Alcohol Dependence Questionnaire (SADQ)), changes in quality of life (using World Health Organizations brief quality of life questionnaire (WHOQOL-BREF)), changes in self-reported treatment effectiveness (using Treatment Effectiveness Assessment (TEA)) and changes in anxiety (using Generalized Anxiety Disorder scale (GAD-7)). Finally, data on the subjective experience of the treatment (using Ego Dissolution Inventory (EDI), Emotional Breakthrough Inventory (EBI) and Mystical Experience Questionnaire (MEQ30)) will be collected and used in a regression model with baseline measures to assess predictors of treatment response on measures of depression and AUD .

ELIGIBILITY:
Please contact the project team for a full and detailed list of inclusion/exclusion criteria

Inclusion Criteria:

* Currently abstinent from alcohol
* At least moderate depression without psychotic features
* Minimum Montgomery-Åsberg Depression Rating Scale (MADRS) of 20
* Alcohol dependence
* Admitted for inpatient addiction therapy at University Hospital of North Norway

Exclusion Criteria:

* Intoxicated or in significant withdrawal from alcohol or drug use
* Not able to give adequate informed consent
* Current or past history of schizophrenia, schizophreniform disorder, paranoid delusional disorder, schizoaffective disorder
* Current or historical diagnosis of schizophrenia in a first degree relative
* Cardiovascular conditions: recent stroke (< 1 year from informed consent), recent myocardial infarction (< 1 year from informed consent), uncontrolled hypertension (>150/100 mm Hg) or recent arrhythmia (< 1 year from informed consent; clinically significant arrhythmia requiring treatment at hospital)
* Liver (Child-Pughs Class C) or kidney (Creatinin clearance < 30 mL/min) failure
* Heart failure (the New York Heart Association Functional Classification (NYHA) class III or IV)
* Chronic respiratory failure (requiring long-term oxygen therapy (LTOT) and/or Global Initiative for Chronic Obstructive Lung Disease system (GOLD) stage 3 or higher)
* Previous anaphylactic reaction to ketamine or midazolam
* Illegal use of ketamine the last 6 months
* Pregnancy or breastfeeding
* Current or suspected increased intracranial pressure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Depression | Within 3 days after final treatment session
  Change from baseline using rater-blinded Montgomery-Åsberg Depression Rating Scale (MADRS) (range 0-60; higher score indicate worse outcome)

SECONDARY OUTCOMES:
Alcohol craving tonic | Repeated measurements from baseline and 1 day, 1 week, 2 weeks and 4 weeks after final treatment session
  Penn Alcohol Craving Scale (PACS) (range 0-30; higher score indicate worse outcome)
Alcohol craving phasic | Repeated measurements from baseline and 1 day, 1 week, 2 weeks and 4 weeks after final treatment session
  Alcohol Craving Questionnaire - Short version (ACQ-short) (range 12-84; higher score indicate worse outcome)
Depression response/remission | Repeated measurements from baseline and 1 day, 1 week, 2 weeks and 4 weeks after final treatment session
  Rates of response (50% or more reduction in MADRS from baseline) and remission (9 points or less in MADRS)
Relapse risk | From baseline until 6 months after baseline
  Incidence of relapse in each group (defined as two or more consecutive heavy drinking days)
Time until relapse | From baseline until 3 and 6 months after baseline
  Average time from final treatment session until relapse

OTHER OUTCOMES:
Duration of antidepressant effect (blinded-rater assessed) | From baseline until 6 months after baseline
  Change in Montgomery-Åsberg Depression Rating Scale (MADRS) (range 0-60; higher score indicate worse outcome)
Duration of antidepressant effect (self-report) | From baseline until 6 months after baseline
  Change in the Beck Depression Inventory-II (BDI-II) (Range 0-63; higher score indicate worse outcome)
Tolerability using the ketamine side effect tool (KSET) | Up to 1 month
  Physician-reported tolerability of each treatment session (good, moderate and poor)
Tolerability using the ketamine side effect tool (KSET) | Up to 1 month
  Patient-reported tolerability of each treatment session (good, moderate and poor)
Cambridge Neuropsychological Test Automated Battery (CANTAB): Stop Signal Task (SST); Spatial Working Memory (SWM) task; Intra-Extra Dimensional Shift (IED) task; Paired Associates Learning (PAL) task; Emotional Bias Task (EBT) | Within 3 days after final treatment session
  Assess within- and between-group changes in neurocognitive function from baseline to within three days from the final treatment session: SST (Range 0-1000; Lower score indicate better outcome); SWM (Range: 2-14; Lower score indicates better outcome); IED (Range: 0-402; Lower score indicates better outcome); PAL (Range: 0-70; Lower score indicates better outcome); EBT (Range: 0-15; Higher score indicates better outcome (more happy))
Adverse reaction frequency | Up to 6 months
  Frequency of adverse reactions
Adverse reaction severity | Up to 6 months
  Number of mild, moderate and severe adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Ole K Grønli, Assoc Prof, Study Director — University Hospital of North Norway; Andreas W Blomkvist, M.D., Principal Investigator — University Hospital of North Norway